CLINICAL TRIAL: NCT06131112
Title: Macrophage PET/CT Imaging for the Diagnosis of Cardiac Sarcoidosis
Brief Title: Macrophage PET/CT Imaging Using 64Cu-DOTATATE for the Diagnosis of Cardiac Sarcoidosis
Acronym: CuDOSIS
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Finn Gustafsson, Professor, Rigshospitalet, Denmark
Other Study IDs: H-23035676
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: 22 patients with clinically suspected cardiac sarcoidosis
  Interventions: Diagnostic Test: 64Cu-DOTATATE PET/CT scan
- Group B: 22 patients with known cardiac sarcoidosis
  Interventions: Diagnostic Test: 64Cu-DOTATATE PET/CT scan
- Group C: Up to 10 patients with clinically suspected or confirmed acute lymphocytic myocarditis
  Interventions: Diagnostic Test: 64Cu-DOTATATE PET/CT scan
- Group D: 22 patients with NET without known inflammatory heart disease who have previously been scanned with 64Cu-DOTATATE PET/CT as part of their routine diagnostic work-up or follow-up (control group)

INTERVENTIONS:
Diagnostic Test: 64Cu-DOTATATE PET/CT scan — Patients in group A-C will have a 64Cu-DOTATATE PET/CT scan performed in addition to routine clinical procedures. Group D has had 64Cu-DOTATATE PET/CT performed as part of their clinical diagnostic work-up or follow-up; these data are retrospectively identified and included in the study, and group D will not be subject to any scans in the study.
  Groups: Group A; Group B; Group C

SUMMARY:
The purpose of the CuDOSIS study is to examine the diagnostic value of activated macrophage imaging in patients with or under evaluation for cardiac sarcoidosis. The PET/CT tracer 64Cu-DOTATATE is used as a tool to identify activated macrophages. The trial is an open-label prospective study. The study will include 54 participants from the Department of Cardiology and the Department of Clinical Physiology, Nuclear Medicine, and PET at Rigshospitalet. Further, the study will include data from 22 patients with NET who have been scanned with 64Cu-DOTATATE PET/CT previously as negative controls.

Participants will be included in the following groups:

Group A: 22 patients with clinically suspected cardiac sarcoidosis Group B: 22 patients with known cardiac sarcoidosis Group C: Up to 10 patients with clinically suspected or confirmed acute lymphocytic myocarditis Group D: 22 patients with NET without known inflammatory heart disease who have previously been scanned with 64Cu-DOTATATE PET/CT as part of their routine diagnostic work-up or follow-up (control group)

DETAILED DESCRIPTION:
Cardiac involvement is considered a serious condition and a frequent cause of death in patients with sarcoidosis. 18F-FDG PET/CT is currently used as part of the diagnostic criteria for cardiac sarcoidosis, but it has shown limitations in the evaluation of cardiac sarcoidosis due to the high physiological uptake of FDG in normal cardiac muscle. Elaborate preparations are required for patients including either a low-carbohydrate diet followed by long fasting or heparin loading before FDG-PET. In heparin loading, the rare adverse effect of heparin-induced thrombocytopenia should be considered. Therefore, it is of interest to find a PET/CT tracer that displays high sensitivity and specificity without requiring thorough patient preparation and minimizing any adverse effects.

A potential tracer is the somatostatin-based tracer 64Cu-DOTATATE, which is routinely used for the diagnosis and monitoring of treatment response in patients with neuroendocrine tumors. Inflammatory cells, including macrophages that are found in sarcoid granulomas, express somatostatin receptors on their surface, whereas normal cardiomyocytes do not. This allows for the potential use of macrophage imaging in cardiac sarcoidosis.

In the CuDOSIS trial, groups A and B (suspected and confirmed cardiac sarcoidosis, respectively) will be scanned with 64Cu-DOTATATE PET/CT in addition to the routinely performed 18F-FDG PET/CT. Further, to examine whether the macrophage infiltration pattern is different in patients with cardiac sarcoidosis and other inflammatory heart diseases, a group of patients with confirmed or clinically suspected myocarditis will be included (group C); this group will only be scanned with 64Cu-DOTATATE PET/CT. Finally, data from a group of patients with neuroendocrine tumours (negative controls) who have previously been scanned with 64Cu-DOTATATE will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age => 18 years
* Group A: 22 patients with clinically suspected cardiac sarcoidosis Group B: 22 patients with known cardiac sarcoidosis Group C: Up to 10 patients with clinically suspected or confirmed acute lymphocytic myocarditis Group D: 22 patients with NET without known inflammatory heart disease who have previously been scanned with 64Cu-DOTATATE PET/CT as part of their routine diagnostic work-up or follow-up (control group)

Exclusion Criteria:

* Severe obesity (weight > 140 kg)
* Pregnancy (negative point-of-care urine/serum human chorion gonadotropin is required in all fertile women)
* Severe claustrophobia
* Known allergy to 64Cu-DOTATATE
* Clinically critical condition which makes PET/CT impossible
* Diabetes with insulin dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adults (18 years or older) from the Department of Cardiology and Department of Clinical Physiology, Nuclear Medicine, and PET at Rigshospitalet. The study will include a total of 76 participants: 54 patients from groups A-C and data from 22 patients from group D.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Tracer uptake - cardiac sarcoidosis and neuroendocrine tumor (negative control) | 2 years
  The proportion of patients with tracer uptake in the heart on 64Cu-DOTATATE PET/CT in patients with verified cardiac sarcoidosis and the proportion of patients without tracer uptake in the heart on 64Cu-DOTATATE PET/CT for patients with a neuroendocrine tumor without a history of inflammatory heart disease (the control group).

SECONDARY OUTCOMES:
24-month rates of adverse outcomes | 2 years
  Death, heart failure hospitalizations, decrease of left ventricular ejection fraction to <10% and <50%, new-onset ventricular tachycardia, new-onset atrioventricular block, implantable cardioverter-defibrillator implantation, shocks from implantable cardioverter-defibrillator, pacemaker implantation, cardiac resyncronization therapy
Tracer uptake - myocarditis | 2 years
  The proportion of patients with tracer uptake in the heart on 64Cu-DOTATATE PET/CT in patients with verified acute lymphocytic myocarditis
Distribution of tracer uptake | 2 years
  The distribution of tracer uptake in the heart in patients with cardiac sarcoidosis and acute lymphocytic myocarditis, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD,PhD,DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The overall results of the trial will be made available. Individual participant data (IPD) will not be made available.